CLINICAL TRIAL: NCT01373229
Title: Lenalidomide in Combination With Plerixafor in Patients With Previously Treated Chronic Lymphocytic Leukemia
Brief Title: Lenalidomide + Plerixafor in Previously Treated Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Collaborators: Celgene Corporation (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00026715; RV0622 (Other: Celgene)
Record Dates: First submitted 2011-06-12; First posted 2011-06-14 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-07

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Chronic Lymphocytic Leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; plerixafor; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide + Plerixafor+ Rituximab (Experimental): 1. Lenalidomide 5mg by mouth (PO) daily beginning cycle 1 day 1.
  2. Stage 1: increase by 2.5mg every 7 days to a maximum dose of 10mg.
  3. Stage 2: plerixafor will be added after 28 days of 10mg dose maintenance and white blood cell count (WBC) <100.0 x 109 / L.
  4. Dose cohorts of escalating subcutaneous (SC) thrice weekly plerixafor with continuous 10mg lenalidomide:
     * Cohort 1: 0.24 mg/kg
     * Cohort 2: 0.32 mg/kg
     * Cohort 3: 0.42 mg/kg
     * Cohort 4: 0.54 mg/kg
  5. Stage 3: Rituximab 375mg/m2 will be added on day 1 of cycles 5-12, day 1 of combination therapy for subjects with PR.
  6. Subjects will then continue single agent lenalidomide until disease progression.
  Interventions: Drug: Lenalidomide + Plerixafor (+ Rituximab)

INTERVENTIONS:
Drug: Lenalidomide + Plerixafor (+ Rituximab) — 1. Lenalidomide 5mg by mouth (PO) daily beginning cycle 1 day 1.
  2. Stage 1: increase by 2.5mg every 7 days to a maximum dose of 10mg.
  3. Stage 2: plerixafor will be added after 28 days of 10mg dose maintenance and white blood cell count (WBC) <100.0 x 109 / L.
  4. Dose cohorts of escalating subcutaneous (SC) thrice weekly plerixafor with continuous 10mg lenalidomide:
     * Cohort 1: 0.24 mg/kg
     * Cohort 2: 0.32 mg/kg
     * Cohort 3: 0.42 mg/kg
     * Cohort 4: 0.54 mg/kg
  5. Stage 3: Rituximab 375mg/m2 will be added on day 1 of cycles 5-12, day 1 of combination therapy for subjects with PR.
  6. Subjects will then continue single agent lenalidomide until disease progression.
  Other Names: Revlimid; Mozobil; Rituxan

SUMMARY:
In research studies, lenalidomide (also called Revlimid) has shown some response in chronic lymphocytic leukemia (CLL); however, responses are usually partial responses that occur after several months of taking the study drug. It is thought that by adding the drug plerixafor (also called Mozobil) responses may be improved and/or occur sooner.

The main purpose of this study is to determine the dose of plerixafor that is safe to use in combination with lenalidomide. The study will also look at the response rates of the combination of lenalidomide and plerixafor and the effect the study drugs have on CLL cells.

DETAILED DESCRIPTION:
The combination of lenalidomide and plerixafor will be evaluated in this single institution, open label clinical study of subjects with relapsed chronic lymphocytic leukemia (CLL). The overall design of the phase 1 study includes up to three treatment "stages."

Each subject will receive lenalidomide 5mg by mouth daily beginning on cycle 1 day 1. If tolerated, the dose will be increased by 2.5mg every 7 days to a maximum dose of 10mg by mouth daily (Stage 1). Once the subject is stably maintained on a daily dose of lenalidomide of 10mg daily and the white blood cell (WBC) count is <100.0 x 109 / L, and has been taking lenalidomide for at least 28 days, plerixafor will be added (Stage 2). In the dose escalation phase, 4 different doses of plerixafor in combination with lenalidomide will be studied in cohorts of 3 to 6 subjects each, following a standard "3 + 3" format:

* Cohort 1: plerixafor 0.24 mg/kg subcutaneous (SC) daily thrice weekly (Mon, Wed, Fri)
* Cohort 2: plerixafor 0.32 mg/kg SC daily thrice weekly (Mon, Wed, Fri)
* Cohort 3: plerixafor 0.42 mg/kg SC daily thrice weekly (Mon, Wed, Fri)
* Cohort 4: plerixafor 0.54 mg/kg SC daily thrice weekly (Mon, Wed, Fri) Plerixafor will be administered for 3 weeks of each cycle (days 1, 3, 5, 8, 10, 12, 15, 17, and 19) followed by a 1 week rest period. Lenalidomide dosing will be continuous.

An interim assessment of response will be performed after 4 cycles of combination therapy:

* Subjects achieving a complete response (CR) by National Cancer Institute (NCI)-96 criteria will continue lenalidomide monotherapy (plerixafor is discontinued) until disease progression.
* Subjects achieving a partial response (PR) will continue both lenalidomide and plerixafor. Additionally, rituximab 375mg/m2 will be added on day 1 of each subsequent cycle beginning with cycle 5, day 1 of combination therapy. (Stage 3). Treatment with the combination of lenalidomide and plerixafor will continue for a maximum of 12 cycles of combination therapy. Subjects may receive up to 8 doses of rituximab concurrent with lenalidomide and plerixafor on day 1 of each cycle. Subjects will then continue single agent lenalidomide until disease progression.
* Subjects with stable disease may continue lenalidomide and plerixafor at the discretion of the investigator and the subject. Rituximab 375 mg/m2 will be added on day 1 of each subsequent cycle. Treatment, dose, schedule, and duration are the same as for subjects achieving a PR.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of chronic lymphocytic leukemia (CLL) or Small lymphocytic lymphoma (SLL) as established by the National Cancer Institute (NCI) Working Group Response Criteria (NCI 96 Criteria).
* Received one or more prior therapies for CLL.
* Subjects must have symptomatic disease requiring therapy as defined by the protocol.
* >/= 4 weeks from prior cancer therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of </= 2.
* All study subjects must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

* Prolymphocytic leukemia (PLL).
* Richter's (large cell) transformation.
* Prior allogeneic transplant within 12 months or prior allogeneic transplant > 12 months currently receiving immunosuppressants.
* Active autoimmune hemolytic anemia.
* Central nervous system (CNS) involvement.
* Chronic enteral corticosteroids > 10mg prednisone or equivalent.
* Evidence of laboratory tumor lysis syndrome (TLS) by Cairo-Bishop Definition of Tumor Lysis Syndrome
* Use of any other experimental drug or therapy within 28 days of baseline
* Major surgery within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Rizzieri, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the CLL clinic at Duke Medical Center from January 2012 to December 2013.
Pre-assignment Details: 21 subjects were consented to this study. Six (6) were screen failures; therefore, only 15 subjects began the treatment regimen which included a lenalidomide run-in phase. Three (3) subjects were unable to complete the run-in phase. Three (3) subjects died prior to completing stage 2, and so were not evaluable for DLT.
Groups:
- Lenalidomide + Plerixafor+ Rituximab: 1. Lenalidomide 5mg by mouth (PO) daily beginning cycle 1 day 1.
  2. Stage 1: increase by 2.5mg every 7 days to a maximum dose of 10mg.
  3. Stage 2: plerixafor will be added after 28 days of 10mg dose maintenance and white blood cell count (WBC) <100.0 x 109 / L.
  4. Dose cohorts of escalating subcutaneous (SC) thrice weekly plerixafor with continuous 10mg lenalidomide:
     * Cohort 1: 0.24 mg/kg
     * Cohort 2: 0.32 mg/kg
  5. Stage 3: Rituximab 375mg/m2 will be added on day 1 of cycles 5-12, day 1 of combination therapy for subjects with PR.
  6. Subjects will then continue single agent lenalidomide until disease progression.
Period: Overall Study
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Started | 15
Completed | 9
Not Completed | 6
Not completed — Death | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Time Frame: 4-16 months
Measure: Number; unit: mg/kg
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Number analyzed (Participants) | 9
mg/kg | 0.24

2. Secondary Outcome: Overall Response (Complete Response/Partial Response)
Description: NCI 96 Response Criteria
  CR (Complete Response):
  Lymphadenopathy = none > 1.5cm Hepatomegaly = none Splenomegaly = none Blood lymphocytes = <4000 per microliter Marrow = normocellular, <30% lymphocytes, no B-lymphoid nodules. Platelet count = >100,000 per microliter Hemoglobin = >11.0 grams per deciliter Neutrophils = >1500 per microliter
  PR (Partial Response):
  Lymphadenopathy = Decrease >/= 50% Hepatomegaly = Decrease >/= 50% Splenomegaly = Decrease >/= 50% Blood lymphocytes = Decrease >/= 50% from baseline Marrow = 50% reduction in marrow infiltrate or B-lymphoid nodules. Platelet count = >100,000 per microliter or increase >/= 50% over baseline Hemoglobin = >11.0 grams per deciliter or increase >/= 50% over baseline Neutrophils = >1500 per microliter or increase >/= 50% over baseline
Time Frame: at the end of 4 months of combination treatment and at 2 months after completion of therapy
Population: Three (3) subjects were unable to complete the run-in phase. Three (3) subjects died prior to completing stage 2, and three (3) subjects were unable to complete 4 cycles of combination therapy. Therefore, only 6 subjects were analyzed for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: time from day 1 of treatment to disease progression, death, or 2 years, whichever comes first
Population: Subjects who experienced disease progression
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Number analyzed (Participants) | 3
months | 11 (1)

4. Secondary Outcome: Overall Survival (OS)
Time Frame: the time from day 1 of treatment to death or 2 years, whichever comes first
Population: Subjects who died on study
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Number analyzed (Participants) | 8
months | 5.5 (10)

5. Secondary Outcome: Reduction in Severity of B Symptoms
Description: Reduction in the severity of the following B symptoms will be assessed: fever ≥ 101F, chills, night sweats, and anorexia with weight loss.
Time Frame: at the end of stage 1 (lenalidomide alone), at the end of stage 2 (4 months of combination), and at 2 months post-completion of therapy
Population: Data were not collected and the Outcome will never be analyzed
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Number analyzed (Participants) | 0

6. Secondary Outcome: Reduction in the Frequency of Blood and Platelet Transfusions
Description: The change in number of transfusions from pre- to post-treatment will be calculated and summarized across all patients by giving the minimum, the 25th, 50th (median) and the 75th percentile and the maximum.
Time Frame: 4 weeks prior to therapy and in the 4 weeks following the completion of therapy
Population: Data were not collected and the Outcome will never be analyzed
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Lenalidomide + Plerixafor+ Rituximab
Serious Adverse Events (participants affected / at risk) | 14/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Plerixafor+ Rituximab (N=15)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide + Plerixafor+ Rituximab (N=15)
Anemia (Blood and lymphatic system disorders) | 13 (14)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 5 (5)
Fatigue (General disorders) | 9 (12)
Fever (General disorders) | 3 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (5)
Pain (General disorders) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 13 (27)
Platelet count decreased (Investigations) | 11 (16)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 2 (4)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2)
Hot flashes (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes